CLINICAL TRIAL: NCT02663700
Title: Dose Escalation Study of Sanaria's Irradiated Sporozoite Vaccine (PFSPZ Vaccine), Followed by a Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of PfSPZ Vaccine in Malaria-Experienced Adults in Burkina Faso
Brief Title: Safety and Immunogenicity of Sanaria's Irradiated Sporozoite Vaccine (PfSPZ Vaccine) in Malaria-Experienced Adults in Burkina Faso
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 15-0001
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07-12

CONDITIONS: Plasmodium Falciparum Infection
Keywords: Adults; Burkina Faso; malaria; PfSPZ Vaccine; Placebo; Randomized
MeSH Terms: conditions — Malaria | interventions — Artesunate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1.8x10^6 sporozoites 2 doses (Experimental): To be completed after safety data from Cohorts 1 and 2 are reviewed. Vaccination with 1.8x10^6 sporozoites on study weeks 3 and 11. n=8
  Interventions: Biological: PfSPZ Vaccine
- 2.7x10^6 sporozoites 2 doses (Experimental): To be completed after safety data from Cohort 3 is reviewed. Vaccination with 1.8x10^6 sporozoites on study weeks 5 and 13. n=8
  Interventions: Biological: PfSPZ Vaccine
- 2.7x10^6 sporozoites 3 doses (Experimental): Subjects to be assigned 1:1 to either PfSPZ vaccine (pending safety data from cohort 4) or placebo. Subjects will be administered the intervention on a 0, 8, and 16 week schedule (study days 1, 57, and 113). n=80
  Interventions: Drug: Artesunate; Biological: PfSPZ Vaccine; Other: Placebo
- 4.5x10^5 sporozoites 2 doses (Experimental): Initial vaccination arm. Vaccination with 4.5x10^5 sporozoites on study weeks 1 and 9. n=8
  Interventions: Biological: PfSPZ Vaccine
- 9x10^5 sporozoites 2 doses (Experimental): Initial vaccination arm. Vaccination with 9x10^5 sporozoites on study weeks 1 and 9. n=8
  Interventions: Biological: PfSPZ Vaccine

INTERVENTIONS:
Drug: Artesunate — Four tablets of 50mg each, totaling 200mg will be given in a single calendar day
  Arms: 2.7x10^6 sporozoites 3 doses
Biological: PfSPZ Vaccine — PfSPZ is a candidate vaccine, it consists of a suspension of purified, live-attenuated cryopreserved Pf sporozoites in a cryoprotectant.
Other: Placebo — Placebo
  Arms: 2.7x10^6 sporozoites 3 doses

SUMMARY:
This study is a phase 1, randomized, double-blind, placebo-controlled, dose escalation trial of Sanaria's irradiated sporozoite vaccine (PfSPZ vaccine). The primary objective of this protocol is to determine the safety and reactogenicity of the PfSPZ Vaccine in malaria-experienced healthy adults. The study duration shall be 34 months and subject participation duration shall be 15-26 months.

DETAILED DESCRIPTION:
This study is a phase 1, randomized, double-blind, placebo-controlled, dose escalation trial of Sanaria's irradiated sporozoite vaccine (PfSPZ vaccine). The primary objective of this study is to determine the safety and reactogenicity of the PfSPZ Vaccine in malaria-experienced healthy adults. The secondary objective is to evaluate vaccine-induced anti-CSP antibody immune responses. The study duration shall be 34 months and subject participation duration shall be 15-26 months.

ELIGIBILITY:
Inclusion Criteria:

1. A male or non-pregnant female aged 21-40 years inclusive at the time of screening.
2. For women, willingness not to become pregnant until 1 month after the last vaccination*.

   *Pre-menopausal female participants will be referred to the local family planning clinic, which offers several means of contraception that are approved and recommended by the Burkina Faso Ministry of Health. Contraception (male or female condoms, diaphragm or cervical cap with spermicide, intrauterine device, or hormone-based contraceptive) should be started 30 days before the first vaccination and continue until 30 days after last vaccination.
3. Written informed consent obtained from the participant before screening.
4. Available and willing to participate in follow-up for the duration of study.
5. Residing in Sapone region and environs.
6. Appear to be in generally good health based on clinical and laboratory investigation.

Exclusion Criteria:

1. Previous vaccination with an investigational malaria vaccine.
2. Use of an investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days before the first study vaccination, or planned use up to 30 days after last vaccination.
3. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months before the first vaccination*.

   *This includes any dose level of oral steroids, but not inhaled steroids or topical steroids.
4. Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first study vaccination with the exception of tetanus toxoid.
5. Confirmed or suspected immunosuppressive or immunodeficient condition.
6. Confirmed or suspected autoimmune disease.
7. History of allergic reactions or anaphylaxis to artesunate and artemisinin derivatives, vaccinations or to any vaccine component.
8. History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care.
9. History of allergy to any component of the vaccine formulation, including human serum albumin.
10. Use or planned use of any drug with anti-malarial activity during the course of the study except for antimalarial medication administered by study clinicians.
11. History of splenectomy.
12. Confirmed or suspected pregnancy or current breastfeeding.
13. Laboratory evidence of liver disease (ALT > / = 1.25 x upper limit of normal).
14. Laboratory evidence of renal disease (serum or plasma creatinine > upper limit of normal).
15. Laboratory evidence of hematologic disease (platelet count <115,000/mm^3, or hemoglobin <11.2 g/dL for males and <9.5 g/dL for females).
16. Seropositive for hepatitis B surface antigen or hepatitis C virus (hepatitis C antibody).
17. Seropositive for HIV.
18. Sickle cell trait carriage or sickle cell disease.
19. Administration of immunoglobulin and/or any blood products within the three months preceding the first study vaccination or planned administration during the study period. 20. Simultaneous participation in any other interventional clinical trial.

21. Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, severe malnutrition, or any other clinical findings that may increase the risk of participating in the study*.

*As determined by the PI. 22. Other condition that in the opinion of the PI would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol. 23. Documented history of non-febrile seizures or atypical (complex) febrile seizures.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Occurrence of Grade 3 unsolicited adverse events (AEs) considered related to vaccination | Day 1 through Day 28
Occurrence of Grade 3 unsolicited adverse events (AEs) considered related to vaccination | Day 57 through Day 83
Occurrence of serious adverse events (SAEs) at any point during the study period | Day 1 through Day 645
Occurrence of serious adverse events (SAEs) considered related to vaccination | Day 1 through Day 28
Occurrence of serious adverse events (SAEs) considered related to vaccination | Day 57 through Day 83
Occurrence of solicited reactions | Day 1 through Day 8
Occurrence of solicited reactions | Day 57 through Day 64

SECONDARY OUTCOMES:
Antibody titers against P. falciparum circumsporozoite protein (CSP) at serology time points | Day 1 through Day 127

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme - Research and Training, Ouagadougou, Kadiogo, Burkina Faso

REFERENCES:
- [Derived] Potter GE, Callier V, Shrestha B, Joshi S, Dwivedi A, Silva JC, Laurens MB, Follmann DA, Deye GA. Can incorporating genotyping data into efficacy estimators improve efficiency of early phase malaria vaccine trials? Malar J. 2023 Dec 19;22(1):383. doi: 10.1186/s12936-023-04802-0. PMID 38115002
- [Derived] Potter GE, Callier V, Shrestha B, Joshi S, Dwivedi A, Silva JC, Laurens MB, Follmann DA, Deye GA. Can incorporating genotyping data into efficacy estimators improve efficiency of early phase malaria vaccine trials? Res Sq [Preprint]. 2023 Sep 22:rs.3.rs-3370731. doi: 10.21203/rs.3.rs-3370731/v1. PMID 37790581